CLINICAL TRIAL: NCT05442905
Title: Quadratus Lumborum Versus Transversus Abdominis Plane Block Versus Caudal Block for Postoperative Analgesia After Pediatric Inguinal Hernia : Double-Blinded Randomized Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mona Mohamed Mogahed, Associate professor, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 35565/6/22
Record Dates: First submitted 2022-06-29; First posted 2022-07-05 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Quadratus Lumborum Block; Transversus Abdominis Plane Block; Caudal Block; Postoperative Pain; Inguinal Hernia
MeSH Terms: conditions — Pain, Postoperative; Hernia, Inguinal | interventions — Propofol; Anesthesia, Intravenous; Atracurium; Sevoflurane

STUDY DESIGN:
Intervention Model Description: Group Q: will receive quadratus lumborum block the patient will be placed in lateral positionGroup T: will receive TAP block with 0.7mL/kg of 0.25% bupivacaine under US guidance. A linear high frequency ultrasound probe (6-13 MHz) will be placed transversely in the mid axillary line between the iliac crest and the costal margin.
  Group C: will receive caudal block with 1mL/kg of 0.25% bupivacaine, with children in left lateral position.
Who Masked: Participant, Outcomes Assessor
Masking Description: The 3 analgesic twchniques were described to the parents preoperatively and they will agree to give their child either of them and To maintain blinding, postoperative evaluation of pain scores will be done by an anesthesiologist, who will be not involved in administering block.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Quadratus lumborum block group (Active Comparator): will receive quadratus lumborum block the patient will be placed in lateral position, the probe will be placed on the crista iliaca anterior superior. After the external oblique, internal oblique, and transversus abdominis muscles will be seen, the probe will be moved to the posterior and the quadratus lumborum muscle will be observed. A 22-gauge, 80 mm insulated Quince-type needle (Uniplex; Pajunk, Geisingen, Germany) will be moved from the anterolateral plane to the posteromedial plane, and confirmation will be made using 0.5 mL/kg saline; after a negative aspiration, 0.7 mL/kg (0.25%) bupivacaine will be applied to the posterior of the quadratus lumborum muscle and the thoracolumbar fascia in between the quadratus lumborum and latissimus dorsi muscles.
  Interventions: Drug: propofol; Drug: Atracurium Besylate; Drug: sevoflurane
- Transversus abdominis block group (Active Comparator): will receive TAP block with 0.7mL/kg of 0.25% bupivacaine under US guidance. A linear high frequency ultrasound probe (6-13 MHz) will be placed transversely in the mid axillary line between the iliac crest and the costal margin. The three layers of muscles, the external oblique, the internal oblique, and the transversus abdominis will be identified. Using the in-plane technique, needle will be inserted (from anterior to posterior direction) until the tip of the needle will reach between the internal oblique and the transversus abdominis. Hydro dissection with 1-2 mL saline will be done to separate the fascial layers. After the correct localization, 20 mL of the drug will beinjected with repeated aspiration to avoid the accidental intravascular injection.
  Interventions: Drug: propofol; Drug: Atracurium Besylate; Drug: sevoflurane
- Caudal block group (Active Comparator): will receive caudal block with 1mL/kg of 0.25% bupivacaine, with children in left lateral position. with all aseptic measures caudal block will be performed using 25 G needle in left lateral decubitus position. Needle position will be confirmed by the pop felt during penetration of the sacrococcygeal ligament, further ensured by doing whoosh test using 0.5 mL of air injection 0.25% bupivacaine 1mL/kg will be administered after negative aspiration of blood and CSF. Intraoperative hemodynamic parameters will be recorded throughout the surgery at fixed intervals (at time of skin incision then after every 5 min till the end of surgery).
  Interventions: Drug: propofol; Drug: Atracurium Besylate; Drug: sevoflurane

INTERVENTIONS:
Drug: propofol — Anesthesia will be induced with propofol 2-3mg/kg
  Other Names: Intravenous anesthesia
Drug: Atracurium Besylate — Atracurium 0.15mg/kg used for muscle relaxation before intubation
  Other Names: Muscle relaxant
Drug: sevoflurane — sevoflurane(1%-2%) used during anesthesia
  Other Names: Inhalational anesthesia

SUMMARY:
Background: Multimodal analgesia (MMA) is the current standard practice to provide postoperative analgesia. The aim of this study is to compare the analgesic efficacy of quadratus lumborum (QL) block versus transversus abdominis plane (TAP) block versus caudal block as an adjunct to MMA.

Methods: In a prospective, randomized, controlled study, 180 children of age 2 8 years and ASA grade Ӏ and ӀӀ, undergoing elective inguinal hernia surgery will be randomly allocated into 3 groups: Group Q (n = 60) will receive USG guided QL block with 0.7mL/kg of 0.25% bupivacaine and Group C (n = 60) will receive caudal block with 1mL/kg of 0.25% bupivacaine and Group T (n = 60) will receive USG guided TAP block with 0.5mL/kg of 0.25% bupivacaine. Postoperatively, all the subjects will be assessed at 2, 4, 6, 8, 12, 18, and 24 hours. The primary outcome will be the time to first analgesic request. The secondary outcomes will be the pain scores during rest and movement, number of doses of morphine, variation in hemodynamic parameters and adverse effects, if any.

DETAILED DESCRIPTION:
This prospective, randomized, comparative study will be conducted at Tanta University Hospitals from August 2022 to March 2023. Total 180 patients of ASA physical status Ӏ ӀӀ, aged 2-8 years, scheduled for inguinal hernia surgery will be randomized into three groups of 60 patients each, using a computer generated random number table. Exclusion criteria will include lack of consent by parents, blood coagulopathies, local infection, vertebral deformity, and allergy to drugs.

Group Q: will receive quadratus lumborum block the patient will be placed in lateral position, the probe will be placed on the crista iliaca anterior superior. After the external oblique, internal oblique, and transversus abdominis muscles will be seen, the probe will be moved to the posterior and the quadratus lumborum muscle will be observed. A 22-gauge, 80 mm insulated Quince-type needle (Uniplex; Pajunk, Geisingen, Germany) will be moved from the anterolateral plane to the posteromedial plane, and confirmation will be made using 0.5 mL/kg saline; after a negative aspiration, 0.7 mL/kg (0.25%) bupivacaine will be applied to the posterior of the quadratus lumborum muscle and the thoracolumbar fascia in between the quadratus lumborum and latissimus dorsi muscles.

Patients in: Group T: will receive TAP block with 0.7mL/kg of 0.25% bupivacaine under US guidance. A linear high frequency ultrasound probe (6-13 MHz) will be placed transversely in the mid axillary line between the iliac crest and the costal margin. The three layers of muscles, the external oblique, the internal oblique, and the transversus abdominis will be identified. Using the in-plane technique, needle will be inserted (from anterior to posterior direction) until the tip of the needle will reach between the internal oblique and the transversus abdominis. Hydro dissection with 1-2 mL saline will be done to separate the fascial layers. After the correct localization, 20 mL of the drug will beinjected with repeated aspiration to avoid the accidental intravascular injection.

Group C: will receive caudal block with 1mL/kg of 0.25% bupivacaine, with children in left lateral position. with all aseptic measures caudal block will be performed using 25 G needle in left lateral decubitus position. Needle position will be confirmed by the pop felt during penetration of the sacrococcygeal ligament, further ensured by doing whoosh test using 0.5 mL of air injection 0.25% bupivacaine 1mL/kg will be administered after negative aspiration of blood and CSF. Intraoperative hemodynamic parameters will be recorded throughout the surgery at fixed intervals (at time of skin incision then after every 5 min till the end of surgery).

All patients will be visited 1 day prior to surgery and will be explained about the anesthesia technique and perioperative course. Each patient will undergo a thorough pre anesthetic check. On arrival in OT, multipara monitoring of ECG, SpO2, NIBP will be established. Base line parameters (SpO2 , pulse rate, SBP, DBP) will be recorded. Patient will be pre medicated with glycopyrrolate 0.005mg/kg, midazolam 0.05mg/kg, and fentanyl 2µg/kg intravenously (IV) through already secured IV line, and ringer lactate infusion will be started. After pre oxygenation with 100% O2 , anesthesia will be induced with propofol 2-3mg/kg and atracurium 0.6mg/kg; endotracheal intubation will be done using appropriate size endotracheal tube. Anesthesia will be maintained with O2 :N2 O ratio 40:60 and sevoflurane(1%-2%) and atracurium 0.15mg/kg SOS. In Group T, patients will be placed in supine position and the abdomen exposed, skin and transducer will be aseptically prepared. The abdominal wall will be scanned using a linear array transducer probe(6-13 MHz) in the multibeam mode, connected to a portable ultrasound unit (S Nerve® SonoSite, Bothell, WA, USA). Probe will be placed in midline over the rectus abdominis muscle at umbilicus level and will be traced laterally to region above the iliac crest to the petit triangle. A 22 G short beveled block needle will be inserted in plane with transducer, in anterior posterior direction. After visualization of needle tip in between internal oblique and transversus abdominis fascial sheath, local anesthetic 0.7mL/kg of bupivacaine 0.25% will be deposited. Correct local anesthetic drug placement will be indicated by hypoechoic elliptical fluid pocket between these two muscles.

To maintain blinding, postoperative evaluation of pain scores will be done by an anesthesiologist, who will be not involved in administering block. Postoperative pain will be assessed by CHEOPS score in which six parameters (cry, facial expression, child verbal, torso, touch, and leg movements) are included. Duration of postoperative analgesia, total number of rescue analgesic requirement and total dose of rescue analgesic required in 24h and any side effects (hypotension, bradycardia, respiratory depression, urinary retention, postoperative nausea and vomiting) will be recorded. Pain scores ≥ 6 for rescue analgesia in form of syrup paracetamol 10mg/kg orally will be administered.

ELIGIBILITY:
Inclusion Criteria:

* patients of ASA physical status Ӏ or ӀӀ
* scheduled for inguinal hernia surgery

Exclusion Criteria:

* lack of consent by parents
* blood coagulopathies.
* local infection.
* vertebral deformity.
* allergy to drugs

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
The time to first analgesic request | 24 hours postoperatively
  The time to first analgesic request is recorded by a nurse unaware about the typy of block.

IPD SHARING:
Plan to Share IPD: Undecided
Authors haven't decided to make individual participant data (IPD) available to other researchers yet.